CLINICAL TRIAL: NCT04472195
Title: Just-In-Time Rapid Cycle Deliberate Practice Simulation Intubation Training Among Novice Pediatric Anesthesia Trainees: A Randomized Control Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Children's Hospital (Other)
Responsible Party: Principal Investigator, Stephen Flynn, Attending Anesthesiologist, Boston Children's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB-P00034169
Record Dates: First submitted 2020-07-08; First posted 2020-07-15 (Actual); Last update posted 2025-01-15 (Actual); Status verified 2025-01

CONDITIONS: Anesthesia

STUDY DESIGN:
Intervention Model Description: Non-crossover, Prospective Randomized Controlled Trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): The experimental group will review a pre-induction airway management plan for their upcoming case and undergo a scripted 10-minute RCDP session with an airway coach within 1 hour of patient intubation. The intubation approach (DL vs. video assisted DL) will be chosen by the primary case attending and communicated to the airway coach to simulate the planned laryngoscopy attempt. The experimental group will then proceed with their scheduled case with a member of the research team observing the laryngoscopy attempt(s) to capture data.
  Interventions: Other: Simulation Airway Coaching
- Control (No Intervention): The trainees in the control group will have no interventions by the research team, only observation of the intubation and documentation of the same details.

INTERVENTIONS:
Other: Simulation Airway Coaching — Airway coaching on laryngoscopy technique for intubation of neonates/infants within 1 hour of case utilizing RCDP simulation technique.
  Arms: Experimental

SUMMARY:
The purpose of this study is to assess the impact of Just-In-Time (J-I-T) Rapid Cycle Deliberate Practice (RCDP) Simulation Training on laryngoscopy competency among novice pediatric anesthesia trainees.

DETAILED DESCRIPTION:
Multiple intubation attempts in infants are potentially more harmful than previously suspected. Emerging literature suggests each additional attempt past an initial laryngoscopy correlates with a two-fold increase in complications. Therefore, striving to secure the neonate/infant airway on the first attempt is optimal for infant safety. Novice trainees lack experience with airway management in small children. To promote a patient safety culture among the multitude of rotating trainees at Boston Children's Hospital the investigators would like to augment airway management with Rapid Cycle Deliberate Practice Simulation Training (RCDP). Rotating trainees at BCH main campus will be prospectively randomized to experimental vs. control group for intubation of neonates and infants less than or equal to 12 months of age. Infants with known congenital heart disease, known or suspected difficult airways, or COVID-19 positive status will be excluded from the study. The experimental group will review a pre-induction airway management plan for their upcoming case and rapid cycle deliberate practice (RCDP) on a simulator with an anesthesia attending coaching on technique prior to real patient intubation. Primary outcome measure will be first attempt success rate. Other outcome measures include: complication rates, a team developed Likert scale that investigates intubation competency and utility of JIT/RCDP training, and NASA-TLX (a validated cognitive task load index).

The study would be the first to directly determine how and if simulation-based pediatric airway interventions are immediately transferable to actual clinical environments in pediatric anesthesiology. Such a study may change how training programs prepare novices for "game time" performance and become a new standard of care in airway management training.

ELIGIBILITY:
Inclusion Criteria:

* Anesthesia Residents
* SRNA
* Pediatric Anesthesia Fellows

Exclusion Criteria:

* Medical Students
* Off-Service Rotators

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 182 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
1st attempt success rate | Through study completion, anticipated 12-15 months
  Trainee first attempt success rate will be observed by the study team

SECONDARY OUTCOMES:
Complication rate | Through study completion, anticipated 12-15 months
  Trainee complication rates of laryngoscopy will be observed by the study team
Self evaluation of neonate/infant laryngoscopy | Through study completion, anticipated 12-15 months
  Trainees will fill out Likert questions developed in conjunction with Boston Children's Survey Methodologist
Evaluation of utility of JIT/RCDP | Through study completion, anticipated 12-15 months
  Trainees will fill out Likert Questions developed in conjunction with Boston Children's Survey Methodologist
Cognitive Load in intubating patient | Through study completion, anticipated 12-15 months
  NASA-TLX will be administered to trainees to evaluate cognitive task load

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Flynn, MD, Principal Investigator — Boston Children's Hospital
Locations (1):
- Boston Children's Hopsital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Galvez JA, Acquah S, Ahumada L, Cai L, Polanski M, Wu L, Simpao AF, Tan JM, Wasey J, Fiadjoe JE. Hypoxemia, Bradycardia, and Multiple Laryngoscopy Attempts during Anesthetic Induction in Infants: A Single-center, Retrospective Study. Anesthesiology. 2019 Oct;131(4):830-839. doi: 10.1097/ALN.0000000000002847. PMID 31335549
- [Background] Park RS, Rattana-Arpa S, Peyton JM, Huang J, Kordun A, Cravero JP, Zurakowski D, Kovatsis PG. Risk of Hypoxemia by Induction Technique Among Infants and Neonates Undergoing Pyloromyotomy. Anesth Analg. 2021 Feb 1;132(2):367-373. doi: 10.1213/ANE.0000000000004344. PMID 31361669
- [Background] Fiadjoe JE, Nishisaki A, Jagannathan N, Hunyady AI, Greenberg RS, Reynolds PI, Matuszczak ME, Rehman MA, Polaner DM, Szmuk P, Nadkarni VM, McGowan FX Jr, Litman RS, Kovatsis PG. Airway management complications in children with difficult tracheal intubation from the Pediatric Difficult Intubation (PeDI) registry: a prospective cohort analysis. Lancet Respir Med. 2016 Jan;4(1):37-48. doi: 10.1016/S2213-2600(15)00508-1. Epub 2015 Dec 17. PMID 26705976
- [Background] Park R, Peyton JM, Fiadjoe JE, Hunyady AI, Kimball T, Zurakowski D, Kovatsis PG; PeDI Collaborative Investigators; PeDI collaborative investigators. The efficacy of GlideScope(R) videolaryngoscopy compared with direct laryngoscopy in children who are difficult to intubate: an analysis from the paediatric difficult intubation registry. Br J Anaesth. 2017 Nov 1;119(5):984-992. doi: 10.1093/bja/aex344. PMID 29028952
- [Background] Else SDN, Kovatsis PG. A Narrative Review of Oxygenation During Pediatric Intubation and Airway Procedures. Anesth Analg. 2020 Apr;130(4):831-840. doi: 10.1213/ANE.0000000000004403. PMID 31567323
- [Background] Hunt EA, Duval-Arnould JM, Nelson-McMillan KL, Bradshaw JH, Diener-West M, Perretta JS, Shilkofski NA. Pediatric resident resuscitation skills improve after "rapid cycle deliberate practice" training. Resuscitation. 2014 Jul;85(7):945-51. doi: 10.1016/j.resuscitation.2014.02.025. Epub 2014 Mar 4. PMID 24607871
- [Background] Ericsson KA. Acquisition and maintenance of medical expertise: a perspective from the expert-performance approach with deliberate practice. Acad Med. 2015 Nov;90(11):1471-86. doi: 10.1097/ACM.0000000000000939. PMID 26375267
- [Background] Ericsson KA and Pool R. Peak: Secrets From the New Science of Expertise. Boston, Mass. Houghton Mifflin Harcourt; 2016.
- [Background] Braga MS, Tyler MD, Rhoads JM, Cacchio MP, Auerbach M, Nishisaki A, Larson RJ. Effect of just-in-time simulation training on provider performance and patient outcomes for clinical procedures: a systematic review. BMJ Simul Technol Enhanc Learn. 2015 Oct 5;1(3):94-102. doi: 10.1136/bmjstel-2015-000058. eCollection 2015. PMID 35515199
- [Background] Kessler D, Pusic M, Chang TP, Fein DM, Grossman D, Mehta R, White M, Jang J, Whitfill T, Auerbach M; INSPIRE LP investigators. Impact of Just-in-Time and Just-in-Place Simulation on Intern Success With Infant Lumbar Puncture. Pediatrics. 2015 May;135(5):e1237-46. doi: 10.1542/peds.2014-1911. Epub 2015 Apr 13. PMID 25869377
- [Background] Nishisaki A, Donoghue AJ, Colborn S, Watson C, Meyer A, Brown CA 3rd, Helfaer MA, Walls RM, Nadkarni VM. Effect of just-in-time simulation training on tracheal intubation procedure safety in the pediatric intensive care unit. Anesthesiology. 2010 Jul;113(1):214-23. doi: 10.1097/ALN.0b013e3181e19bf2. PMID 20526179
- [Derived] Flynn SG, Park RS, Jena AB, Staffa SJ, Kim SY, Clarke JD, Pham IV, Lukovits KE, Huang SX, Sideridis GD, Bernier RS, Fiadjoe JE, Weinstock PH, Peyton JM, Stein ML, Kovatsis PG. Coaching inexperienced clinicians before a high stakes medical procedure: randomized clinical trial. BMJ. 2024 Dec 16;387:e080924. doi: 10.1136/bmj-2024-080924. PMID 39681397